CLINICAL TRIAL: NCT03116529
Title: Neoadjuvant Anti-PD-L1 (Durvalumab/MEDI4736) Plus Anti-CTLA-4 (Tremelimumab) and Radiation for High Risk Soft-Tissue Sarcoma
Brief Title: Neoadjuvant Durvalumab and Tremelimumab Plus Radiation for High Risk Soft-Tissue Sarcoma
Acronym: NEXIS
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Limited Accrual
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: AstraZeneca (Industry); University of Arizona (Other); West Penn Allegheny Health System (Other)
Responsible Party: Principal Investigator, Vincent Ng, Assistant Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00073356
Record Dates: First submitted 2017-04-12; First posted 2017-04-17 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Soft Tissue Sarcoma
Keywords: Neoadjuvant; Soft Tissue Sarcoma; Immunotherapy; Checkpoint Inhibitor; PD-1 (Programmed Cell Death Protein 1); PD-L1 (Programmed Death Ligand 1); CTLA-4 (Cytotoxic T-Lymphocyte-Associated Protein 4); Radiotherapy; Durvalumab; Tremelimumab; Surgery; Radiation; Combined; Preoperative
MeSH Terms: conditions — Sarcoma; Parkinson Disease 4, Autosomal Dominant Lewy Body; Diabetes Mellitus, Insulin-Dependent, 12 | interventions — Immunotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Neoadjuvant Radiation plus Durvalumab and Tremelimumab Wide Surgical Resection Adjuvant Durvalumab
  Interventions: Combination Product: Combination Radiation, Immunotherapy, Surgery

INTERVENTIONS:
Combination Product: Combination Radiation, Immunotherapy, Surgery — Three doses of Durvalumab (1500 mg) and Tremelimumab (75 mg) given intravenously once every four weeks during radiotherapy prior to surgery.
  Radiation therapy delivered with a minimum dose of 50 Gy and 1.8-2 Gy per fraction. Bulky sarcomas, defined as >10 cms in greatest dimension, receive a single 15 Gy fraction of high-dose spatially fractionated (GRID) radiation therapy within 1-3 days prior to radiation therapy
  Surgical resection is performed at least 5-8 weeks after cessation of radiotherapy and 4 weeks after completion of neoadjuvant immunotherapy.
  Patients with no evidence of disease following surgical resection receive four additional doses and patients with evidence of disease receive nine additional doses of Durvalumab (1500 mg IV) once every four weeks unless there is clear progression of disease.

SUMMARY:
Chemotherapy is controversial for soft tissue sarcoma that has not yet metastasized. Surgery and radiation are effective for local control, but there are no highly effective interventions to prevent metastatic spread of soft tissue sarcoma. Immunotherapy has shown promise in other types of cancer. Combining two types of immunotherapy agents with preoperative radiation may help the immune system recognize the sarcoma and stimulate an anti-tumor immune response.

DETAILED DESCRIPTION:
The main purposes of this study are to evaluate the safety, tolerability, and efficacy of Durvalumab and Tremelimumab in combination with radiation prior to surgical resection of high-risk soft tissue sarcoma in the pelvis and extremities.

Patients will receive the same radiation therapy and surgical care they would receive normally and with no change in timing or duration of each treatment. They will also receive two immunotherapy agents, Durvalumab and Tremelimumab, during radiation prior to surgery, and a single agent, Durvalumab, after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Willingness and ability to comply with the protocol for the duration of the study
* Histologically confirmed intermediate or high grade adult-type soft tissue sarcoma
* Location of tumor is trunk (non-retroperitoneal) or extremities
* Tumor at least 5 cm in greatest dimension and deep to fascia, or locally recurrent, or metastatic, or have had prior inadequate resections
* Judged as at least marginally resectable
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Adequate normal organ and marrow function
* Female subjects must be either of non-reproductive potential (i.e., post-menopausal by history: ≥60 years old and no menses for ≥1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry.
* Females of childbearing potential who are sexually active with a non-sterilized male partner and non-sterilized male subjects who are sexually active with a female partner of childbearing potential must be willing to use 2 methods of effective contraception from time of screening through 180 days after receipt of the final dose of Durvalumab + Tremelimumab combination therapy or 90 days after receipt of the final dose of Durvalumab Monotherapy, whichever is the longer time period.

Exclusion Criteria:

* Primarily bone-based sarcomas that can occur in the soft tissue such as: extra-skeletal Ewing sarcoma, extra-skeletal osteosarcoma, peripheral chordoma, extra-skeletal myxoid chondrosarcoma, and mesenchymal chondrosarcoma
* Predominantly low-grade soft tissue sarcoma, such as solitary fibrous tumor / hemangiopericytoma, well-differentiated liposarcoma, dermatofibrosarcoma protuberans, Kaposi's sarcoma
* Pediatric-type soft tissue sarcoma, such as rhabdomyosarcoma
* Gastrointestinal stromal tumors (GIST)
* Retroperitoneal soft tissue sarcoma
* Patients with extra-pulmonary metastases aside from lymph node involvement
* Surgically unresectable primary lesion
* Symptomatic or uncontrolled brain metastases requiring concurrent treatment, inclusive of but not limited to surgery, radiation and/or corticosteroids.
* Any previous treatment with an anti-PD-1 (programmed cell death protein-1), anti-PD-L1 (programmed death ligand 1) or anti-CTLA-4 (cytotoxic T-lymphocyte-associated protein 4) therapy, including Durvalumab and Tremelimumab
* History of hypersensitivity to Durvalumab or any excipient
* History of hypersensitivity to Tremelimumab or any excipient
* History of hypersensitivity to the combination or comparator agent
* History or clinically confirmed pneumonitis or interstitial lung disease
* Receipt of the last dose of anti-cancer therapy (cytotoxic chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) ≤ 28 days prior to the first dose of study drug (28 days prior to the first dose of study drug for subjects who have received prior TKIs (tyrosine kinase inhibitors) [e.g., erlotinib, gefitinib and crizotinib] and within 6 weeks for nitrosourea or mitomycin C [If sufficient wash-out time has not occurred due to the schedule or PK properties of an agent, a longer wash-out period may be required])
* Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab or tremelimumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid
* Any unresolved toxicity (>grade 2) from previous anti-cancer therapy. NOTE: Subjects with irreversible toxicity that is not reasonably expected to be exacerbated by the investigational product may be included (e.g., hearing loss, peripherally neuropathy)
* Any prior immune-related adverse event (irAE) ≥ Grade 2 while receiving any previous immunotherapy agent, or any unresolved irAE > Grade 1
* Active or prior documented autoimmune disease within the past 2 years. NOTE: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
* History of primary immunodeficiency
* History of allogeneic organ transplant (e.g. solid organ/bone marrow transplant patients)
* Uncontrolled intercurrent illness including, but not limited to:
* Ongoing or active infections
* Cardiac conditions, such as:
* symptomatic congestive heart failure
* uncontrolled hypertension
* unstable angina pectoris
* cardiac arrhythmia
* Active peptic ulcer disease or gastritis
* History of inflammatory bowel disease, ulcerative colitis or Crohn's Disease
* Active bleeding diatheses
* Any subject known to have evidence of acute or chronic hepatitis B or hepatitis C
* Any subject known to have evidence of human immunodeficiency virus (HIV) or acquired immune deficiency syndrome (AIDS)
* Uncontrolled seizures
* Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Fredericia's Correction
* Known history of current or recent clinical diagnosis of tuberculosis (within three months prior to enrollment)
* Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
* Any signs or symptoms of bowel obstruction within 28 days prior to study entry
* History of leptomeningeal carcinomatosis
* Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab or tremelimumab, or active infection
* History of psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
* Previously enrolled in the present study
* Participation in another clinical study with an investigational product during the last 6 months
* Previously enrolled in the present study
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 180 days after the last dose of durvalumab + tremelimumab combination therapy or 90 days after the last dose of durvalumab monotherapy, whichever is the longer time period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
Toxicity: Number of subjects experiencing high-grade toxicity | 90 days after receipt of final dose of Durvalumab monotherapy or 180 days after receipt of final dose of combination Durvalumab/Tremelimumab, whichever is longer
  Number of subjects experiencing high-grade toxicity
Histopathologic Response | At time of surgery
  Number of subjects with an excellent response on histopathologic examination of the surgically removed tumor

SECONDARY OUTCOMES:
Overall Survival Rate | Two years after start of treatment
  Percentage of patients still alive
Overall Survival Rate | Five years after start of treatment
  Percentage of patients still alive
Disease-Specific Survival Rate | Two years after start of treatment
  Percentage of patients who have not died from soft tissue sarcoma
Disease-Specific Survival Rate | Five years after start of treatment
  Percentage of patients who have not died from soft tissue sarcoma
Relapse-Free Survival Rate | Two years after start of treatment
  Percentage of patients who have not had a documented relapse of local or distant disease
Relapse-Free Survival Rate | Five years after start of treatment
  Percentage of patients who have not had a documented relapse of local or distant disease
Radiologic Response To Treatment | At time of surgery
  Best overall response to Neoadjuvant Radiation and Immunotherapy using Response Evaluation Criteria in Solid Tumors (RECIST)
Radiologic Response To Treatment | At time of surgery
  Best overall response to Neoadjuvant Radiation and Immunotherapy using immune-related response criteria (irRC)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Y. Ng, MD, Principal Investigator — University of Maryland Medical Center, Greenebaum Comprehensive Cancer Center
Locations (3):
- United States (3):
  - University of Arizona, Tucson, Arizona
  - University of Maryland Medical Center, Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Allegheny General Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ng VY, Sahlani MN, Fogel JD, Chiu AK, Kallen ME, Davis D, Snider J, Regine W, Bentzen SM, Sausville E. Results of an Integrated Phase I/II Prospective Clinical Trial (NEXIS) for Neoadjuvant Anti-PD-L1 (Durvalumab) and Anti-CTLA-4 (Tremelimumab) With Radiation for High-Risk Soft-Tissue Sarcoma of the Trunk and Extremities. Cureus. 2024 Oct 22;16(10):e72119. doi: 10.7759/cureus.72119. eCollection 2024 Oct. PMID 39575028
- [Derived] Vatner R, James CD, Sathiaseelan V, Bondra KM, Kalapurakal JA, Houghton PJ. Radiation therapy and molecular-targeted agents in preclinical testing for immunotherapy, brain tumors, and sarcomas: Opportunities and challenges. Pediatr Blood Cancer. 2021 May;68 Suppl 2:e28439. doi: 10.1002/pbc.28439. Epub 2020 Aug 22. PMID 32827353
- See also: The Bone Cancer and Soft Tissue Sarcoma Service at Greenebaum Comprehensive Cancer Center at the University of Maryland Medical Center — https://www.umms.org/umgccc/cancer-services/cancer-types/bone-soft-tissue/team